CLINICAL TRIAL: NCT00154453
Title: Age-Related Changes in Myosin Heavy Chain Composition in Human Orbicularis Oculi Muscle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9261701166
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2003-10

CONDITIONS: Aging
Keywords: Aging; Orbicularis oculi; Blepharoplasty; Myosin heavy chain (MHC)

INTERVENTIONS:
Procedure: obtain surgical specimen for analysis

SUMMARY:
Orbicularis oculi muscle is a key structure in the peri-orbital anatomy and is responsible for the major changes of aging in this area. Peri-orbital rejuvenation has been an issue of great interest in plastic surgery. We believe that understanding the age-related histomorphometric changes in orbicularis oculi muscle is important for improving the current rejuvenation techniques or developing the new ones. Nevertheless, a study focusing on this topic has never been performed before, simply because it is difficult and dangerous to perform needle biopsy on orbicularis oculi muscle.

DETAILED DESCRIPTION:
Hundreds of people came to our hospital requesting upper blepharoplasty every year. Taking advantage of the discarded soft tissue in the blepharoplasty surgery, samples of bilateral orbicularis oculi muscle can be easily obtained from patients of various ages. This study is designed to objectively evaluate the age-related changes in human orbicularis oculi muscle by analyzing the composition of isoforms of myosin heavy chain (MHC), which is the predominant protein in skeletal muscle. MHC isoforms exist in different types of muscle fibers, and determines the maximum contraction speed of the muscle fiber. Therefore, The composition of MHC isoforms represents the composition of different types of muscle fiber.

These muscle specimens are stored with liquid nitrogen right after surgery. In the lab, the specimens are sectioned to 40μm in thickness, and soaked in special buffer solution. After electrophoresis and staining, bands of different types of MHC can be visualized. The gel is scanned and processed with an image analysis system. The density of each band can be determined, and the ratio of the different types of MHC can be calculated.

By dividing the subjects who had their orbicularis oculi muscle sampled during upper blepharoplasty operation into age groups of 20, 30, 40, 50, 60 and 70 years, these MHC subtypes composition ratios can be compared among the different groups. Therefore, the age-related changes of the composition of different muscle types can be concluded.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving blepharoplasty

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-01; Study Completion 2004-08

PRIMARY OUTCOMES:
Differentiation capability of preadipocyte

SECONDARY OUTCOMES:
Proliferation capability of preadipocyte

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Bih Tang, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital